CLINICAL TRIAL: NCT04344249
Title: Prospective Multicenter Cohort of Patients With Inflammatory Bowel Disease Treated by Infliximab or Vedolizumab During COVID-19 Pandemic
Brief Title: Cohort of Patients With Inflammatory Bowel Disease During COVID-19 Pandemic
Acronym: IBD-COVID-19
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC20_0150
Record Dates: First submitted 2020-04-08; First posted 2020-04-14 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: IBD; COVID
Keywords: IBD; Ulcerative colitis; SARS-CoV-2; infliximab; vedolizumab; Crohn's disease
MeSH Terms: conditions — Colitis, Ulcerative; Crohn Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Multicenter cohort of patients followed for 6 months during the pandemic in France with biocollection of sera and peripheral blood mononuclear cells

DETAILED DESCRIPTION:
Multicenter cohort of patients followed for 6 months during the pandemic in France with biocollection of sera and peripheral blood mononuclear cellsNo data has been published concerning the incidence and prevalence of SARS-CoV-2 infection in patients with IBD and treated by IV infusion of infliximab or vedolizumab. It seems that biotherapies have a minimal impact on the severity of the viral infection but data are scarce. The objectives of the cohort are to quantify the incidence and the prevalence of SARS-CoV-2 in this population of patients, to determine clinical, demographic and biological factors associated with the risk of infection and the severity of the disease with a Multicenter cohort of patients followed for 6 months during the pandemic in France with biocollection of sera and peripheral blood mononuclear cells.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (>18 years), know Crohn's disease or ulcerative colitis, treated by infliximab or vedolizumab

Exclusion Criteria:

* not affiliated to a sanitary social insurance

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: all adult patients with Crohn's disease or ulcerative colitis treated by infliximab or vedolizumab
Sampling Method: Non-Probability Sample
Enrollment: 1109 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2021-02-18 (Actual); Study Completion 2021-02-18 (Actual)

PRIMARY OUTCOMES:
IgG and IgM anti SARS-CoV-2 | through study completion, an average of 2 year
  Impact of antibodies du to immunosuppressive protocol on the risk of viral infection

SECONDARY OUTCOMES:
Clinical factors and severity of COVID-19 infection | through study completion, an average of 2 year
  Describe clinical factors of the population of IBD patients treated with vedolizumab or infliximab who develop asymptomatic, pauci-symptomatic non-hospitalized and severe IBD requiring hospital management.
  * weight (Kg)
  * height (m)
  * ABO Group ....
demographic factors and severity of COVID-19 infection | through study completion, an average of 2 year
  Describe demographic factors of the population of IBD patients treated with vedolizumab or infliximab who develop asymptomatic, pauci-symptomatic non-hospitalized and severe IBD requiring hospital management.
  * ACCOMMODATION
  * HOUSING AREA
  * number of people at home ....
pharmacologic factors and severity of COVID-19 infection | through study completion, an average of 2 year
  Describe residual rates of treatments (edolizumab or infliximab) of the population of IBD patients who develop asymptomatic, pauci-symptomatic non-hospitalized and severe IBD requiring hospital management.

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Nantes, Nantes, France